CLINICAL TRIAL: NCT04671836
Title: Lorazepam Effects on Neuroimaging Measures: A Pilot Study
Brief Title: Lorazepam Effects on Neuroimaging Measures
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No longer interested in conducing study
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Juan Gallego Angel, Assistant Investigator, Northwell Health
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20-0773
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Lorazepam; Neuroimaging
Keywords: lorazepam; functional connectivity; spectroscopy; healthy volunteers
MeSH Terms: interventions — Lorazepam; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lorazepam first (Experimental): This arm comprises of participants who were randomized to receive lorazepam 1 mg prior to the first MRI scan and then placebo on the second MRI scan a week later.
  Interventions: Drug: Lorazepam 1Mg Tablet; Drug: Placebo
- Placebo first (Placebo Comparator): This arm comprises of participants who were randomized to receive placebo prior to the first MRI scan and then lorazepam 1 mg orally prior to the second MRI scan a week later.
  Interventions: Drug: Lorazepam 1Mg Tablet; Drug: Placebo

INTERVENTIONS:
Drug: Lorazepam 1Mg Tablet — 1 mg, white, five-sided (shield shape) tablet with a raised "A" on one side and "BPI" and "64" impressed on scored reverse side. NDC 0187-0064-01 - Bottles of 100 tablets; NDC 0187-0064-50 - Bottles of 500 tablets; NDC 0187-0064-10 - Bottles of 1000 tablets.
  The pharmacy at the Zucker Hillside Hospital will encapsulate both lorazepam 1 mg and placebo pills to make them look the same. On the day of the scan, the research coordinator or the PI will pick up the blinded study medication (lorazepam or placebo) and will administer it to the participant. One hour later, the participant will be placed in the scanner to complete the MRI.
Drug: Placebo — Placebo will be purchased and encapsulated by the pharmacy at the Zucker Hillside Hospital.

SUMMARY:
This within-subject, double blind, randomized controlled study will investigate the effects of a widely used benzodiazepine (BZD), lorazepam, on various neuroimaging measures. The investigators will be assessing the relationship of lorazepam to resting state functional connectivity and other neuroimaging measures. Specifically, the investigators will be using a pre-identified metric, the striatal connectivity index (SCI), (Sarpal et al. 2015, 2016), a prognostic biomarker of treatment response assessing the connectivity between regions of the striatum and the cortex. The investigators hypothesize that lorazepam administration will be associated with greater SCI values compared with placebo administration; consistent with previous work suggesting short-acting benzodiazepines increase functional connectivity across brain networks.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18-40
4. In general good health as evidenced by medical history
5. Ability to take oral medication and be willing to adhere to the study medication regimen
6. For women of reproductive potential, negative pregnancy test and agreement to use a medically accepted birth control method.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy or lactation
2. Contraindications to MR imaging (i.e. pacemaker)
3. Known allergic reactions to components of the lorazepam
4. Current smoker or tobacco use
5. Concurrent use of any psychotropic medications, anticonvulsants, opioids or any other medication with effects on the CNS.
6. Acute narrow-angle glaucoma
7. Current or past history of a substance use disorder and/or a positive urine toxicology test.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
To understand the impact of lorazepam on functional connectivity measures collected using resting state functional magnetic imaging (rs-fMRI). | 2 weeks
  SCI, a parameter that captures the connectivity between the stratum and the cortex, is a primary candidate for a prognostic biomarker that may guide individual treatment. Exploratory functional connectivity analyses between other brain regions will be conducted as well.

SECONDARY OUTCOMES:
The goal is to study the impact of lorazepam on glutamate, glutamine and GABA in the striatum. | 2 weeks
  Metabolite concentrations measured in parts per million (ppm) for Glutamate, glutamine and GABA; obtained with Magnetic Resonance Spectroscopy (MRS).

CONTACTS AND LOCATIONS:
Overall Officials: Juan A Gallego, MD, Principal Investigator — Northwell Health
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sarpal DK, Argyelan M, Robinson DG, Szeszko PR, Karlsgodt KH, John M, Weissman N, Gallego JA, Kane JM, Lencz T, Malhotra AK. Baseline Striatal Functional Connectivity as a Predictor of Response to Antipsychotic Drug Treatment. Am J Psychiatry. 2016 Jan;173(1):69-77. doi: 10.1176/appi.ajp.2015.14121571. Epub 2015 Aug 28. PMID 26315980
- [Result] Sarpal DK, Robinson DG, Lencz T, Argyelan M, Ikuta T, Karlsgodt K, Gallego JA, Kane JM, Szeszko PR, Malhotra AK. Antipsychotic treatment and functional connectivity of the striatum in first-episode schizophrenia. JAMA Psychiatry. 2015 Jan;72(1):5-13. doi: 10.1001/jamapsychiatry.2014.1734. PMID 25372846